CLINICAL TRIAL: NCT03307941
Title: Assessment of Metabolic and Pathological Response to Treatment With RCT and ImT Before Surgery in Locally Advanced Esophageal and Gastro-esophageal Junction Cancer: ARTemIS-Eso, a Three-level, Open-label, Phase I-II Study
Brief Title: Assessment of Metabolic & Path Response w/ RCT & ImT Before Surgery in Locally Advanced Esoph and Gastro-esoph Jction CA
Acronym: ARTEMIS-Eso
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Suspended collaboration with the company providing the study drug
Sponsor: Jules Bordet Institute (Other)
Collaborators: Innate Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IJB-GASTON-002-ARTEMIS-Eso; 2016-000935-42 (EudraCT Number)
Record Dates: First submitted 2016-10-27; First posted 2017-10-12 (Actual); Last update posted 2017-12-19 (Actual); Status verified 2017-12

CONDITIONS: Adenocarcinoma of the Esophagus; Adenocarcinoma of the Gastroesophageal Junction; Squamous Cell Carcinoma of the Esophagus
MeSH Terms: conditions — Adenocarcinoma Of Esophagus; Esophageal Squamous Cell Carcinoma | interventions — monalizumab; Oxaliplatin; Fluorouracil; Metabolic Networks and Pathways; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (classic 3+3 design) (Other)
  Interventions: Drug: Monalizumab; Drug: Oxaliplatin; Drug: 5-Fluorouracil; Radiation: Metabolic; Other: Metabolic; Procedure: Surgery

INTERVENTIONS:
Drug: Monalizumab — Monalizumab (IPH2201) is given at the recommended dose of 10 mg/kg, intravenously (infusion during 60 minutes) every two weeks
  Other Names: IPH2201
Drug: Oxaliplatin — A total of 4 cycles of FOLFOX is administrated every 2 weeks with one cycle 15 days prior to the radiotherapy and 3 cycles during the radiotherapy whatever the level
Drug: 5-Fluorouracil — A total of 4 cycles of FOLFOX is administrated every 2 weeks with one cycle 15 days prior to the radiotherapy and 3 cycles during the radiotherapy whatever the level
Radiation: Metabolic — Radiation therapy must start the first day of FOLFOX chemotherapy. Radiation is given once daily for 5 consecutive days; on the days that the patient receives chemotherapy (and monalizumab when applicable), chemotherapy (and monalizumab) should be given prior to radiotherapy.
Other: Metabolic — 18-FDG-PET scan will be performed just before the beginning of radio-chemotherapy (D10-D14) and will be blinded for investigators and patients. Another 18-FDG-PET will be performed before surgery (surgery Day-5 to surgery Day -1) to exclude metastatic evolution
  Other Names: FDG-PET
Procedure: Surgery — Surgery is performed preferably 8 weeks after the completion of the radio-chemotherapy, and it should not be performed less than one week after the last dose of monalizumab

SUMMARY:
ARTemIS-Eso is a phase I-II, three-level, open-label trial with a dose-expansion cohort at recommended schedule in both esophageal cancer histological groups (squamous cell carcinoma and adenocarcinoma) of RCT and ImT administered prior to surgery.

DETAILED DESCRIPTION:
This study is indicated to patients with adenocarcinomas of the esophagus or gastro-esophageal junction and squamous cell carcinoma of the esophagus.

The study consists of 2 parts:

Phase I of the study is composed of the 3 following levels, corresponding to changes in the schedule and the number of administrations of monalizumab:

Level 1: monalizumab (ImT) administration starts 2 weeks after the end of RCT (Total of 3 ImT doses). A maximum of 7 days delay is allowed.

Level 2: monalizumab administration starts directly at the end of RCT (Total of 4 ImT doses). The first dose of monalizumab should be given on the following working day after the last radiotherapy administration.

Level 3: monalizumab administration starts 2 weeks after the start of RCT (total of 6 ImT doses). A maximum of 7 days delay is allowed.

Phase II (Expansion cohort): At the recommended level determined in phase I and according to the number of patients already accrued, approximately 48-51 additional patients (half-SCC and half-ADC) are included with the aim of assessing the activity of the recommended combination.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old
2. ECOG performance status ≤ 1
3. Female and Male
4. Must have histologically confirmed esophageal ADC or SCC or gastro-esophageal junction ADC (Siewert I and II) eligible for a curative intent resection (recommended exploration by EUS and diagnostic laparoscopy in gastro-esophageal junctions) without restriction in age and sex and candidate for neoadjuvant RCT.
5. At least classified clinical T3Nx or any T, N+ according to cTNM version 7.
6. Negative serum pregnancy test (for women of childbearing potential) within 7 (+/-1) days prior to the beginning of treatment.
7. Women of childbearing potential must agree to use one highly effective method of contraception at study entry (if this is not already the case, put in place within 1 week after ICF signature, and at the very latest before 1st administration of study treatment), during the study treatment administration and at least 5 months after the last administration of study treatment.
8. Men must agree to use condom during the course of this study and for at least 5 months after the last administration of the study treatment.
9. Adequate bone marrow function as defined below:

   * Absolute neutrophil count ≥1500/µL or 1.5x109/L
   * Hemoglobin ≥ 9 g/dL
   * Platelets ≥100000/µL or 100x109/L
10. Adequate liver function as defined below:

    * Serum total bilirubin ≤ 1.5 x ULN. In case of known Gilbert's syndrome < 3xUNL is allowed
    * AST (SGOT)/ALT (SGPT) ≤ 2.5 x ULN
    * Alkaline phosphatase ≤ 2.5 x ULN
11. Adequate renal function as defined:

    * Creatinine ≤ 1.5 x UNL or creatinine clearance >60 mL/min
12. Participants must have normal cardiac and pulmonary functions defined with ultrasonography (LVEF>50%) and pulmonary function tests (including DLCO (diffusing capacity factor of the lung for carbon monoxide)).
13. Completion of all necessary screening procedures within 28 days prior to enrolment.
14. Accessible tumour for biopsies through upper gastro-intestinal endoscopy (for translational research activities).
15. Signed Informed Consent form (ICF) obtained prior to any study related procedure and study treatment.
16. For the phase II expansion cohort only, significant FDG uptake at the primary tumour on baseline PET/CT, performed not more than 7 days before the beginning of the first course of CT, defined as SUVmax > 2x the mean liver uptake.

Exclusion Criteria:

Subjects meeting one of the following criteria are not eligible for this study:

1. Patient ineligible for curative intent surgery:

   * T4 with involvement of mediastinal structures as tracheobronchial, recurrent nerve, aorta over 90° of its circumference, vertebral body
   * Tumour ≥ 4cm in diameter developed above the carina
   * Visceral metastasis
   * Metastatic lymph nodes: supraclavicular and/or lombo-aortic
   * Cervical esophageal cancer defined as a tumor involving the lower border of the cricoid cartilage (at the level of the sixth cervical vertebra) to the thoracic inlet 5cm down under, generally between 18 and 20 cm from the dental arcade
2. Uncontrolled concurrent illness or any significant disease that, in the investigator's opinion, would exclude the patient from the study.
3. Absolute contraindication for surgery: respiratory failure (VEMS < 1000mL), weight loss> 20%, renal failure: creatinine > 1.5 ULN, myocardial infarct < 6 months, evolutive cardiopathy, ECOG 3 and 4, non-compensated cirrhosis.
4. Pregnant and/or lactating women.
5. Uncontrolled diabetes.
6. Individuals with a history of a different malignancy within the last 5 years are ineligible except cervical cancer in situ, and early stage basal cell or squamous cell carcinoma of the skin.
7. Patients with active, known or suspected autoimmune disease or condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive systemic treatment.

   * (Exception: patients with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring immunosuppressive systemic treatment, or conditions not expected to recur in the absence of an external trigger, are permitted to be enrolled.
   * Inhaled or topical steroids and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active/autoimmune disease.
8. Patients with diseases known for hypersensitivity to radiotherapy.
9. Prior treatment for esophageal cancer: surgery, radiotherapy, chemotherapy or immunotherapy (in particular but not limited to anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or immune checkpoint pathways, including prior therapy with anti-tumour vaccines or other immuno-stimulatory anti-tumour agents.
10. Positive test for hepatitis B virus surface antigen (HBsAg) or hepatitis C virus (ribonucleic acid or HCV antibody) indicating acute or chronic infection.
11. Positive test for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS).
12. History of allergy to study drug components or excipients.
13. Subject with a significant medical, neuro-psychiatric, or surgical condition, currently uncontrolled by treatment, which, in the principal investigator's opinion, may interfere with completion of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-07-20 (Actual); Primary Completion 2017-12-11 (Actual); Study Completion 2017-12-11 (Actual)

PRIMARY OUTCOMES:
Phase I: determine the feasibility to administer monalizumab | From date of randomization until the date of first documented disease recurrence, assessed up to 28 months
  Successful and safe administration of the combination of radio-chemotherapy and at least 2 doses of immunotherapy
Phase II: pCR rate | At date of surgery, assessed at 16 weeks post randomization
  Defined by the absence of any tumoral cells on the surgical specimen post esophagectomy

SECONDARY OUTCOMES:
Phase I: pCR rate | At date of surgery, assessed at 16 weeks post randomization
  Defined by the absence of any tumoral cells on the surgical specimen post esophagectomy
Phase I: DFS and OS at 2 years after surgery | From date of randomization until the date of first documented event, assessed up to 28 months
  DFS and OS at 2 years after surgery
Phase I: Human Anti-Human Antibodies against monalizumab (HAHA) in serum | Week 5 to 3 months post surgery
  Human Anti-Human Antibodies against monalizumab (HAHA) in serum
Phase II: Two year-disease free survival (DFS) and two year-overall survival (OS) | 2 years after the date the last patient had his surgery provided the trial objectives have been met
  Two year-disease free survival (DFS) and two year-overall survival (OS)
Phase II: Toxicity profile according to CTCAE v.4.03 | From date of randomization until the date of first documented event, assessed up to 28 months
  Toxicity profile according to CTCAE v.4.03
Phase II: Metabolic response after 1 course of CT and before surgery | from week 1 up to the time of surgery
  Metabolic response after 1 course of CT and before surgery
Phase II: Number of the tumour-infiltrating lymphocytes (TILs) | at baseline, after 1 course of CT at week 3 and after surgery at 16 weeks
  Number of the tumour-infiltrating lymphocytes (TILs)

CONTACTS AND LOCATIONS:
Overall Officials: Amelie Deleporte, Physician, Study Chair — Jules Bordet Institute
Locations (1):
- Institut Jules Bordet, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No